CLINICAL TRIAL: NCT03128437
Title: The Relationship Between Anxiety, Mood, and Health Behaviors in Young Adults
Brief Title: Anxiety, Mood, and Health Behaviors in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HM20009285
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Anxiety Sensitivity
Keywords: Anxiety; Young Adults; Health Behaviors
MeSH Terms: conditions — Anxiety Disorders; Health Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Condition (Experimental): 6 aerobic exercise exposures will be completed over the course of 2 weeks.
  Interventions: Behavioral: Aerobic Exercise
- Assessment Only Condition (No Intervention): Participants randomly assigned to the control condition will complete assessments at the same time intervals as the active condition, but will not participate in exercise sessions.
  Assessments will take place at baseline, week 2, week 4, and week 8.

INTERVENTIONS:
Behavioral: Aerobic Exercise — At each of the six exposure sessions, participants will be invited to engage in 2-minute warm-up on the treadmill. Following this warm-up period, participants will be asked to briskly walk or jog on the treadmill at a speed that maintains their heart rate at 60-80% of maximum age-predicted heart rate for 20 minutes using the formula: (220-age) x (0.60 [lower bound] or 0.80 [upper bound]). Participants will be fitted with a heart rate monitor, which will be checked by a research assistant at 5-minute intervals in order to ensure adherence to this prescription; participants will be asked to adjust treadmill speed in order to remain in this range. Following each 20-minute exposure, participants will complete 5 minutes of cool down walking on the treadmill. Assessments will take place at baseline, week 2 (post-intervention), week 4, and week 8.
  Arms: Aerobic Exercise Condition

SUMMARY:
This is a randomized control trial to test the effect of an anxiety sensitivity intervention on health behaviors among 18-35 year-olds.

DETAILED DESCRIPTION:
This is a 2-arm randomized control trial to test the effect of an anxiety sensitivity intervention on health behaviors among 18-35 year-olds. Participants will be 18-35 year-olds with high anxiety sensitivity randomized to 1)Exercise Exposure Intervention or 2)Assessment Only Control Condition. Participants in both groups will be followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35
* Elevated anxiety sensitivity (ASI-3 score >=23)
* Able to safely participate in moderate-intensity physical activity as assessed by the Physical Activity Readiness Questionnaire (PAR-Q), which will be administered during screening

Exclusion Criteria:

* Current aerobic exercise routine - Measured using the L-CAT with an established cut point of >2 (assessed at screening)
* Receiving ongoing psychotherapy or counseling (Self-report at screening)
* Recent change in psychotropic medication for anxiety (Self-report at screening)
* Psychiatric hospitalization in past 6 months (Self-report at screening)
* Current pregnancy (Self-report at screening)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Anxiety sensitivity | 4 weeks
  Anxiety sensitivity represents an individual-level propensity to appraise the experience of anxiety as aversive in terms of social, physical, and/or cognitive consequences. It has been implicated in the maintenance of fear behavior (i.e., avoidance) and the development of clinically significant symptomatology with respect to anxiety and depression. Anxiety sensitivity will be assessed using the Anxiety Sensitivity Index-3.

SECONDARY OUTCOMES:
Physical activity | 4 & 8 weeks
  Physical activity will be assessed using the 7-day Physical Activity Recall questionnaire.
Anxiety sensitivity | 8 weeks
  Anxiety sensitivity represents an individual-level propensity to appraise the experience of anxiety as aversive in terms of social, physical, and/or cognitive consequences. It has been implicated in the maintenance of fear behavior (i.e., avoidance) and the development of clinically significant symptomatology with respect to anxiety and depression. Anxiety sensitivity will be assessed using the Anxiety Sensitivity Index-3.
Heart rate variability | 2 weeks
  A continuous 3 lead ECG (SE-1010 PC ECG, Edan USA) will be acquired for 5 minutes while the subject rests in a supine position in a quiet, private room.
Alcohol use | 4 & 8 weeks
  Quantity and frequency of alcohol use will be assessed using the Timeline Follow-back method (Alcohol TLFB; Sobell & Sobell, 1992). This semi-structured interview asks participants to retrace their behavior and activities over a given timespan in order to assess daily alcohol use.
Binge eating | 4 & 8 weeks
  Consistent with methods reported in Deboer et al., (2012), binge eating frequency will be assessed continuously using item 8 of the Eating Disorder Diagnostic Scale (EDDS; Stice, Telch, & Rizvi, 2000): "How many times have you eaten an unusually large amount of food and experienced a loss of control?" This question will be integrated into the semi-structured interview procedures as described above in order to increase accuracy of responses.
Sleep | 4 & 8 weeks
  The Insomnia Severity Index (ISI; Bastien, Vallieres, & Morin, 2001) will also be administered in order to capture more nuanced information about participants' sleep quality. Seven items assessing severity of insomnia symptoms comprise the ISI, with higher scores indicating more significant sleep disturbances.
Exercise Stage of Change | 4 & 8 Weeks
  Stage of exercise behavior change will be measured using a 6-item self-report questionnaire developed by Marcus, Selby, Niaura, & Rossi (1992). Participants respond to each item using a 5-point Likert scale ranging from "strongly disagree" to "strongly agree."

CONTACTS AND LOCATIONS:
Overall Officials: Jessica LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, School of Medicine, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanoye A, Rybarczyk B, Evans R, Leahey T, LaRose J. Pilot randomized clinical trial targeting anxiety sensitivity: effects on physical activity. Cogn Behav Ther. 2022 May;51(3):257-271. doi: 10.1080/16506073.2021.1954082. Epub 2021 Aug 10. PMID 34374633